CLINICAL TRIAL: NCT04943471
Title: Assessment of Personality Traits in Patients With Symptomatic Floaters Seeking Consultation for Its Treatment
Brief Title: Personality Traits in Patients Seeking a Consultation for Treatment for Floaters
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 301344
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Myodesopia
MeSH Terms: interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients will be given a questionnaire: All patients will be given the Big Five Questionnaire
  Interventions: Other: Big Five Questionnaire, Patient health questionnaire-9 and generalised anxiety disorder -7 questionnaire

INTERVENTIONS:
Other: Big Five Questionnaire, Patient health questionnaire-9 and generalised anxiety disorder -7 questionnaire — Questionnaire

SUMMARY:
This study aims to assess if certain personality traits are move prevalent in patients seeking consultation for treatment of floaters, despite good visual acuity and no other ocular pathology compared to the normal population.

DETAILED DESCRIPTION:
This study aims to assess if certain personality traits are move prevalent in patients seeking consultation for treatment of floaters, despite good visual acuity and no other ocular pathology compared to the normal population. A questionnaire utilising a validated personality trait assessment the 'Big Five Inventory' will collect information patients who have sought a consultation (or already had treatment in the form of vitrectomy) for floaters. We will also assess whether these patients are suffering from any degree of depression or anxiety using two validated screening questionnaires; the patient health questionnaire-9 to screen for depression, and the generalised anxiety disorder - 7 questionnaire to screen for anxiety. Identifying personality traits of patients who seek further help and potential therapeutic intervention, could help clinicians identify the individual factors that lead to this debilitating condition in some patients, despite having a healthy eye and may help determine future non-surgical minimally-interventional therapeutic approaches in the future

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged 18 or over who have contacted an Ophthalmologist for a consultation for treatment for myodesopsia which has lasted for over 3 months

Exclusion Criteria:

* • Patients with co-existing ocular pathology e.g. uveitis, glaucoma, pathological myopia (refractive error > -6D)

  * Patients with cognitive impairment or learning difficulties that would affect their ability to access and complete the questionnaire
  * Patients with known personality disorders
  * Patients must be able to read, speak and understand English so they can comprehend the patient information sheet and questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 or over who have contacted an Ophthlamologist for a consultation for treatment for myodesopia which has lasted more than 3 months
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Degree of neuroticism in patient group compared to an established normative database | 6 months
  Patients will complete a big five inventory questionnaire. This assesses five personality traits using a likert scale. There are 44 statements. The degree to which patients agree with each statement calculates their score, with certain statements being reversed scored. Patients indicate agreement by stating they either disagree strongly, disagree a little, neither agree nor disagree, agree a little or strongly agree. In items scored normally disagree strongly will give the minimum score of 1, with strongly agreeing giving a score of 5. For items which are reversed scored disagree strongly will give a score of 5, and strongly agreeing will give a score of 1.

SECONDARY OUTCOMES:
Difference in degree of other 4 personality measures in the big five inventory and normative database | 6 months
  The difference in extraversion, agreeableness, conscientiousness, openness in the recruited patient database and normative database will be analysed
Difference in degree of anxiety and depression between normative database and recruited patients | 6 months
  The patient health questionnaire -9 and generalised anxiety disorder questionnaire will be given to patients. These are commonly used tools to screen/assess depression and anxiety. With both questionnaires the higher the score, the greater the degree of anxiety or depression. The frequency of depression and anxiety within the patient group will be assessed and multivariate regression analysis will be done to see if there is an association with any of the personality traits.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided